CLINICAL TRIAL: NCT00001521
Title: An Open, Randomized, Long-Term Clinical Trial of Flutamide, Testolactone, and Reduced Hydrocortisone Dose vs. Conventional Treatment of Children With Congenital Adrenal Hyperplasia
Brief Title: Three Drug Combination Therapy Versus Conventional Treatment of Children With Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960033; 96-CH-0033
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-05-08

CONDITIONS: Congenital Adrenal Hyperplasia (CAH)
Keywords: Congenital Adrenal Hyperplasia (CAH); Intervention; Children
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Fludrocortisone; Hydrocortisone; Letrozole; Flutamide; Testolactone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational therapy (Experimental): Children with congenital adrenal hyperplasia (CAH) and bone ages of 2-13 years in boys and 2-11 years in girls were randomized to receive antiandrogen (flutamide 10mg/kg/day orally), aromatase inhibitor (testolactone - 20mg/ kg/day orally OR letrozole - 1.5mg/m^2 body surface area orally), low-dose hydrocortisone (6-8 mg/m^2/day orally), and fludrocortisone (100-200 mcg/day, depending on lab evaluation, orally). Participants received the four-drug regimen until the age of 13 in the girls and 14 in the boys and then were switched to standard therapy. Female participants on investigational drugs were continued on flutamide until attainment of final adult height or two years post menarche. Participants who experienced early puberty received GnRH agonist therapy: depot leuprolide 7.5-15 mg/kg monthly intramuscularly or deslorelin 4 mcg/kg/day (adjusted based on weight and response) subcutaneously.
  Interventions: Drug: Fludrocortisone; Drug: Hydrocortisone; Drug: Letrozole; Drug: Flutamide; Drug: Testolactone
- Standard therapy (Experimental): Children with congenital adrenal hyperplasia (CAH) and bone ages of 2-13 years in boys and 2-11 years in girls received standard therapy/conventional treatment (with hydrocortisone and fludrocortisone). Participants received hydrocortisone approximately 10-15 mg/m^2/day orally, not exceeding 25mg/m^2/day, and fludrocortisone 100-200 mcg/day orally depending on lab evaluation. Participants who experienced early puberty received GnRH agonist therapy: depot leuprolide 7.5-15 mg/kg monthly intramuscularly or deslorelin 4 mcg/kg/day (adjusted based on weight and response) subcutaneously.
  Interventions: Drug: Fludrocortisone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Fludrocortisone — Mineralocorticoid needed to replace aldosterone deficiency. Patients will continue to receive an optimal fludrocortisone dose
Drug: Hydrocortisone — Glucocorticoid needed to replace cortisol deficiency. Reduced hydrocortisone dose might normalize the growth and adult stature of children with congenital adrenal hyperplasia
Drug: Letrozole — Aromatase inhibitors work by inhibiting the action of the enzyme aromatase, which converts androgens into estrogens by a process called aromatization.
  Arms: Investigational therapy
Drug: Flutamide — Non steroidal anti-androgen that prevents the action of androgens by blocking receptor sites in target tissue. It may also produce changes in testosterone and estradiol
  Arms: Investigational therapy
Drug: Testolactone — Aromatase inhibitors work by inhibiting the action of the enzyme aromatase, which converts androgens into estrogens by a process called aromatization.
  Arms: Investigational therapy

SUMMARY:
This study was developed to determine if a combination of four drugs (flutamide, testolactone, reduced hydrocortisone dose, and fludrocortisone) can normalize growth in children with congenital adrenal hyperplasia.

The study will take 60 children, boys and girls, and divide them into 2 groups based on the medications given. Group one will receive the new four-drug combination. Group two will receive the standard treatment for congenital adrenal hyperplasia (hydrocortisone and fludrocortisone).

The boys in group one will take the medication until the age of 14 at which time they will stop taking the four-drug combination and begin receiving the standard treatment for congenital adrenal hyperplasia. Girls in group one will take the four-drug combination until the age of 13, at which time they will stop and begin receiving the standard treatment for congenital adrenal hyperplasia plus flutamide. Flutamide will be given to the girls until two years after their first menstrual period or until adult height.

All of the children will be followed until they reach their final adult height. The effectiveness of the treatment will be determined by measuring the patient's adult height.

DETAILED DESCRIPTION:
To test the hypothesis that the regimen of flutamide (an antiandrogen), testolactone or letrozole (an inhibitor of androgen-to-estrogen conversion), and reduced hydrocortisone dose can normalize the growth and adult stature of children with congenital adrenal hyperplasia, and can avoid the complications of supraphysiologic glucocorticoid dosage, 60 children with this disorder will be randomized to receive either the above regimen or conventional treatment until they have reached age 13 years in a girl or age 14 in a boy. After these ages boys will receive the conventional treatment and girls will receive conventional treatment plus flutamide. In girls, flutamide will be continued until 6 months after menarche. All children will be followed until they have attained final adult height. The principal outcome measure will be adult height.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be boys with bone ages 2 to 13 years and girls with bone ages 2 to 11 years with CAH due to classic 21-hydroxylase deficiency.

Subjects must either not yet have undergone pubertal activation of the hypothalamic-pituitary-gonadal axis, or, if pubertal activation has occurred, must be receiving a GnRH agonist to suppress secondary central precocious puberty.

Children with a bone age of 1 to 2 years may enroll in the protocol for optimization of conventional therapy, but will not be randomized to a study arm until the bone age reaches 2.

EXCLUSION CRITERIA:

Children who have concurrent illnesses requiring glucocorticoid treatment (such as severe asthma), or requiring drugs that markedly alter hydrocortisone metabolism (such as anticonvulsants), and children who cannot be brought into reasonable control with conventional treatment (an unusual occurrence).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 1995-06-08 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data is being used for secondary analyses.

REFERENCES:
- [Result] Merke DP, Mallappa A, Parker M, Sukin C, Kulkarni SE, Keil MF, Van Ryzin C, Hill SC, Reynolds JC, Cutler GB Jr, Sinaii N. Adult Height Following Prepubertal Treatment With Antiandrogen, Aromatase Inhibitor, and Reduced Hydrocortisone in CAH. J Clin Endocrinol Metab. 2025 Jun 17;110(7):e2171-e2182. doi: 10.1210/clinem/dgae824. PMID 39672600
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1996-CH-0033.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 participants were consented, two participants withdrew prior to randomization and two were compassionate exemption so were not randomized.
Period: Overall Study
Arm/Group | Investigational Therapy | Standard Therapy
Started | 31 | 31
Moved From Investigational to Standard Therapy | 4 | 0
Completed | 21 | 24
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Noncompliant | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Therapy | Standard Therapy | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 31 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 18 | 21 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 28 | 56
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Adult Height Relative to General Population
Description: Adult height expressed in standard deviation score (SDS) units relative to the general population, with attainment of adult height defined as incremental growth < 1.5 cm over 12 months. Adult height SDS was based on National Health and Nutrition Examination Survey (Centers for Disease Control and Prevention, National Center for Health Statistics) data at 20 years old.
Time Frame: Followed to attainment of adult height, average of 11 years from date of randomization
Population: Modified intention-to-treat population, includes patients who were reassigned from investigational to standard therapy due to drug intolerance.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 27
Standard Deviation Score (SDS) units | -0.34 (0.93) | -0.6 (0.89)

2. Secondary Outcome: Adult Height Relative to Mid-parental Height
Description: Adult height expressed in standard deviation score (SDS) units relative to the mid-parental height for the general population. Adult height is defined as incremental growth < 1.5 cm over 12 months. Adult height SDS was based on National Health and Nutrition Examination Survey (Centers for Disease Control and Prevention, National Center for Health Statistics) data at 20 years old. Mid-parental height was calculated based on reported parental heights calculated as (father's height (cm) + mother's height (cm))/ 2 ± 6.5 (cm).
Time Frame: Followed to attainment of adult height, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 27
Standard Deviation Score (SDS) units
  Overall Participants | -0.45 (0.85) | -0.83 (0.78)
  Males: number analyzed (Participants) | 9 | 17
  Males | -0.89 (0.75) | -0.93 (0.78)
  Females: number analyzed (Participants) | 9 | 10
  Females | -0.02 (0.72) | -0.67 (0.79)

3. Secondary Outcome: Predicted Adult Height
Description: Predicted adult height was calculated using the bone age at the baseline visit or the first available bone age, using the Bayley-Pinneau method. Predicted adult height was calculated as the standard deviation score (SDS) units relative to the general population based on the National Health and Nutrition Examination Survey data (Centers for Disease Control and Prevention (CDC), National Center for Health Statistics) at 20 years old. Baseline was defined as time of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys).
Time Frame: At date of randomization and at pubertal onset (average of seven years from date of randomization)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 25 | 33
Standard Deviation Score (SDS) units
  Baseline | -2.0 (1.5) | -2.1 (1.5)
  Pubertal onset: number analyzed (Participants) | 20 | 31
  Pubertal onset | -0.46 (0.97) | -0.98 (1.01)

4. Secondary Outcome: Predicted Adult Height Change
Description: Changes in predicted adult height from baseline to pubertal onset, pubertal onset to final visit, and baseline to final visit. Adult height standard deviation score (SDS) was based on National Health and Nutrition Examination Survey (Centers for Disease Control and Prevention, National Center for Health Statistics) data at 20 years old. Predicted adult height at baseline was calculated using the bone age at the baseline visit or the first available bone age according to the Bayley-Pinneau method. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: From date of randomization to pubertal onset visit (which on average was seven years), pubertal onset to final visit (average was 4 years), and date of randomization to final visit (average of 11 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 26
Standard Deviation Score (SDS) units
  Baseline to pubertal onset visit | 1.93 (1.29) | 1.10 (1.32)
  Pubertal onset to final visit: number analyzed (Participants) | 16 | 25
  Pubertal onset to final visit | -0.10 (0.66) | 0.14 (0.54)
  Baseline to final visit: number analyzed (Participants) | 17 | 24
  Baseline to final visit | 1.64 (1.23) | 1.20 (1.27)

5. Secondary Outcome: Number of Years Bone Age Remained Unchanged
Description: Number of prepubertal and pubertal years bone age remained unchanged. Baseline bone age was calculated using the bone age at the baseline visit or the first available bone age according to the Bayley-Pinneau method. Change in bone age from baseline to pubertal onset and pubertal onset to final visit was measured in years. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: From date of randomization to pubertal onset visit (which on average was seven years) and pubertal onset to final visit (average was 4 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 27
Years
  Baseline to pubertal onset visit | 3.86 (2.13) | 2.78 (2.43)
  Pubertal onset to final visit | 0.39 (0.68) | 0.70 (0.73)

6. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Changes in body mass index (BMI) were evaluated from baseline to puberty onset and puberty onset to final visit. BMI calculation was based on average of three early morning height measurements by stadiometer and weight measurement by scale for each timepoints. BMI was calculated as the standard deviation score (SDS) units relative to the general population based on the National Health and Nutrition Examination Survey data (Centers for Disease Control and Prevention (CDC), National Center for Health Statistics) at 20 years old. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was time at attainment of adult height, defined as incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
Standard Deviation Score (SDS) units
  Baseline to pubertal onset visit | 0.12 (0.7) | 0.36 (0.79)
  Pubertal onset to final visit: number analyzed (Participants) | 18 | 27
  Pubertal onset to final visit | -0.06 (0.54) | -0.20 (0.61)

7. Secondary Outcome: Body Mass Index (BMI)
Description: Body mass index (BMI) was calculated based on average of three early morning height measurements by stadiometer and weight measurement by scale. BMI was calculated as the standard deviation score (SDS) units relative to the general population based on the National Health and Nutrition Examination Survey data (Centers for Disease Control and Prevention (CDC), National Center for Health Statistics) at 20 years old. Measures evaluated at pubertal onset and at final visit. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: Pubertal onset visit (average of seven years from date of randomization) and at final visit (average of 11 years from date of randomization)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
Standard Deviation Score (SDS) units
  Pubertal onset visit | 1.07 (1.30) | 1.09 (0.93)
  Final visit: number analyzed (Participants) | 18 | 27
  Final visit | 0.79 (1.13) | 0.89 (0.83)

8. Secondary Outcome: Average Annual Growth Velocity
Description: Average annual growth (height) velocity, measured as the change in height over time relative to the population mean and adjusted for age and sex. Measured during the study period from baseline visit to pubertal onset visit (visits occurring approximately every 6 months) and from pubertal onset to adult height. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS) units
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
Standard Deviation Score (SDS) units
  Baseline to pubertal onset | -1.01 (1.84) | -0.34 (2.18)
  Pubertal onset to adult height: number analyzed (Participants) | 18 | 27
  Pubertal onset to adult height | 0.65 (1.42) | -0.29 (1.34)

9. Secondary Outcome: Dose of Oral Hydrocortisone
Description: Dose of oral hydrocortisone participant was taking adjusted for body surface area. Dose was recorded at baseline (first visit), pubertal onset, and at adult height (final visit). Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: At date of randomization, pubertal onset (average of seven years from date of randomization), and at final visit (average of 11 years from date of randomization)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/m2 /day
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 27 | 35
mg/m2 /day
  Baseline | 14.7 (3.8) | 13.9 (3.5)
  Pubertal onset: number analyzed (Participants) | 21 | 31
  Pubertal onset | 7.6 (1.5) | 15.0 (3.6)
  Adult height: number analyzed (Participants) | 18 | 27
  Adult height | 16.4 (3.1) | 16.8 (2.9)

10. Secondary Outcome: Average Daily Dose of Oral Hydrocortisone
Description: Average daily dose of oral hydrocortisone adjusted for body surface area. Dose was measured by developmental periods and for differences between sexes. Doses recorded at every visit, approximately every 6 months. Average dose measured from baseline to pubertal onset, from pubertal onset visit to adult height (final visit), and from baseline to adult height. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/m2 /day
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
mg/m2 /day
  Baseline to adult height: number analyzed (Participants) | 18 | 27
  Baseline to adult height | 10.1 (1.7) | 15.0 (2.4)
  Baseline to pubertal onset: Male: number analyzed (Participants) | 12 | 20
  Baseline to pubertal onset: Male | 9.5 (1.6) | 15.0 (2.8)
  Baseline to pubertal onset: Female: number analyzed (Participants) | 9 | 11
  Baseline to pubertal onset: Female | 9.1 (1.5) | 13.9 (2.6)
  Pubertal onset to adult height: Male: number analyzed (Participants) | 9 | 17
  Pubertal onset to adult height: Male | 14.7 (0.9) | 15.5 (2.5)
  Pubertal onset to adult height: Female: number analyzed (Participants) | 9 | 10
  Pubertal onset to adult height: Female | 9.5 (2.2) | 15.5 (3.0)

11. Secondary Outcome: Percent of Visits With 17-hydroxyprogesterone in the Optimal Range (<1,200 ng/dL)
Description: Percentage of visits where early morning (pre-medication) 17-hydroxyprogesterone measurements fell within the optimal range (<1,200 ng/dL) during the study period from baseline to pubertal onset and pubertal onset visit to final visit, with visits occurring approximately every 6 months. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of visits
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
Percentage of visits
  Baseline to pubertal onset | 11.8 [5.9 to 22.7] | 35.9 [19.4 to 65.2]
  Pubertal onset to adult height: number analyzed (Participants) | 18 | 27
  Pubertal onset to adult height | 0 [0 to 30.0] | 28.6 [11.8 to 54.5]

12. Secondary Outcome: Percent of Visits With Androstenedione in Normal Range
Description: Percentage of visits where early morning (pre-medication) androstenedione measurements fell within the normal range based on age and sex-specific ranges during the study period. Measurements done from baseline to pubertal onset visit, and from pubertal onset visit to adult height (final visit), with visits occurring approximately every 6 months. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage of visits
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
Percentage of visits
  Baseline to pubertal onset | 0 [0 to 10.5] | 45 [28.6 to 78.6]
  Pubertal onset to final visit: number analyzed (Participants) | 18 | 27
  Pubertal onset to final visit | 20.2 [0 to 50.0] | 50.0 [25.0 to 81.8]

13. Secondary Outcome: Average Testosterone
Description: Average testosterone based on early morning (pre-medication) testosterone levels measured for participants approximately every six months. Average testosterone measured from baseline to pubertal onset and from pubertal onset visit to adult height (final visit) by sex. Baseline was defined as date of randomization. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 21 | 31
ng/dL
  Baseline to pubertal onset | 86.3 [42.2 to 100.0] | 24.5 [19.7 to 36.8]
  Pubertal onset to final visit: Males: number analyzed (Participants) | 9 | 17
  Pubertal onset to final visit: Males | 336.0 [303.3 to 492.5] | 418.4 [349.6 to 504.4]
  Pubertal onset to final visit: Females: number analyzed (Participants) | 9 | 10
  Pubertal onset to final visit: Females | 42.3 [33.5 to 155.9] | 34.4 [20.6 to 52.1]

14. Secondary Outcome: Number of Participants With Onset of Early Central Puberty
Description: Number of participants with onset of early central puberty, defined as testicular volume ≥ 4 mL in males before age 10, and breast Tanner stage 2 in females before age 9.
Time Frame: Measured from date of randomization to onset of early central puberty
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 16 | 24
Participants | 12 | 9

15. Secondary Outcome: Average Age at Menarche
Description: Average age at menarche (years) in female participants only.
Time Frame: Followed from date of randomization to onset of menarche
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 9 | 11
Years | 14.7 (1.7) | 13.6 (0.9)

16. Secondary Outcome: Number of Female Participants With Normal Menstrual Cyclicity at Final Visit
Description: Number of female participants with normal menstrual cyclicity at final visit. Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: Measured at single time point at final visit, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 8 | 10
Participants | 4 | 7

17. Secondary Outcome: Number of Participants With Insulin Resistance Based on Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) > 2.5
Description: Number of participants with Insulin resistance based on Homeostasis model assessment of insulin resistance (HOMA-IR) > 2.5 at the final visit. Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: Final visit, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 26
Participants | 8 | 12

18. Secondary Outcome: Average (Median) Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostasis model assessment of insulin resistance (HOMA-IR), a measure of insulin resistance, measured as insulin (μU/mL) × glucose (mmol/L)/22.5 at final visit. HOMA-IR value ≤ 2.5 is considered normal. HOMA-RI value > 2.5 is considered abnormal. Higher HOMA-IR value indicates greater insulin resistance. Final visit was attainment of adult, defined as height with incremental growth <1.5 cm over 12 months.
Time Frame: Measured at single time point at final visit, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 26
Units on a scale | 2.42 [2.12 to 4.82] | 2.29 [1.68 to 3.2]

19. Secondary Outcome: Number of Male Participants With Testicular Adrenal Rest Tumors (TART)
Description: Number of male participants with testicular adrenal rest tumors (TART), measured by scrotal ultrasound, at pubertal onset visit and final visit. Pubertal onset was defined as when patients entered puberty (Tanner 2 breast in females, testicle size ≥ 4 mL in males) or completed therapy with either aromatase inhibitor and/or GnRHa (age 13 years in girls and 14 years in boys). Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 12 | 20
Participants
  Pubertal onset | 4 | 3
  Final visit: number analyzed (Participants) | 9 | 17
  Final visit | 7 | 7

20. Secondary Outcome: Anterior Posterior Spine Bone Mineral Density (BMD) at Final Visit
Description: Anterior posterior spine bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DEXA) scan at final visit. The instrument specific comparisons (in standard deviations) were made to the average peak bone mass of a normal population, i.e. to the average bone mass of persons of the same age and sex as the patient. Final visit is defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: Final visit, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z Scores
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 27
Z Scores | -0.19 (1.28) | -0.25 (0.84)

21. Secondary Outcome: Femoral Neck Bone Mineral Density (BMD) at Final Visit
Description: Femoral neck bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DEXA) scan at final visit. The instrument specific comparisons (in standard deviations) were made to the average peak bone mass of a normal population, i.e. to the average bone mass of persons of the same age and sex as the patient. Final visit was defined as attainment of adult height with incremental growth < 1.5 cm over 12 months.
Time Frame: Final visit, average of 11 years from date of randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z Scores
Arm/Group | Investigational Therapy | Standard Therapy
Number analyzed (Participants) | 18 | 27
Z Scores | -0.07 (1.23) | -0.32 (1.03)

ADVERSE EVENTS:
Time Frame: Up to 16 years from start of study
Description: Reporting for standard therapy included four participants who transition from Investigational to Standard Therapy due to drug intolerance
Arm/Group | Investigational Therapy | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/31 | 10/35
Other Adverse Events (participants affected / at risk) | 31/31 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Therapy (N=31) | Standard Therapy (N=35)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hypoglycaemic seizure (Endocrine disorders) | 0 | 1
Appendicitis (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 8
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Therapy (N=31) | Standard Therapy (N=35)
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 21 | 18
Animal bite (Injury, poisoning and procedural complications) | 0 | 2
Liver function test increased (Investigations) | 6 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 14 | 10
Headache (Nervous system disorders) | 1 | 2
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Somnambulism (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Laceration (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1
Child abuse (Social circumstances) | 1 | 0
Limb reconstructive surgery (Surgical and medical procedures) | 1 | 0
Suture insertion (Surgical and medical procedures) | 2 | 4
Tonsillectomy (Surgical and medical procedures) | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 1
Lip injury (Gastrointestinal disorders) | 1 | 0
Mumps (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Ear infection (Ear and labyrinth disorders) | 11 | 6
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
External ear inflammation (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 30 | 29
Mononucleosis syndrome (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 3 | 0
Genital injury (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Multiple fractures (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 3 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaesthesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Kidney infection (Renal and urinary disorders) | 1 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Nail avulsion (Skin and subcutaneous tissue disorders) | 0 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 0
Varicella (Skin and subcutaneous tissue disorders) | 1 | 1
Bladder training (Surgical and medical procedures) | 0 | 1
Dental care (Surgical and medical procedures) | 0 | 1
Dental operation (Surgical and medical procedures) | 2 | 0
Emergency care (Surgical and medical procedures) | 8 | 10
Female genital operation (Surgical and medical procedures) | 0 | 1
Ligament operation (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT00001521/Prot_SAP_000.pdf